CLINICAL TRIAL: NCT01105130
Title: A Randomized Phase II Dose Finding Study of ArginMax for Its Effect on Erectile Function and Quality of Life in Survivors of Prostate Cancer Previously Treated With Radiotherapy
Brief Title: L-Arginine Supplementation With or Without Enzyme Inhibitors Treating Erectile Function of Prostate Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB00012793; U10CA081851 (NIH); REBACCCWFU 98110 (Other: NCI)
Record Dates: First submitted 2010-04-14; First posted 2010-04-16 (Estimated); Results first posted 2015-07-21 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Male Erectile Disorder; Prostate Cancer; Radiation Toxicity
Keywords: radiation toxicity; male erectile disorder; prostate cancer
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Neoplasms; Radiation Injuries | interventions — Arginine; ArginMax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I - Placebo (Placebo Comparator): Patients receive oral placebo twice daily (total of 6 capsules per day).
  Interventions: Other: Placebo
- Arm II - low dose (Experimental): Patients receive oral L-arginine and oral placebo twice daily (total of 3 capsules of each per day).
  Interventions: Other: Placebo; Drug: Oral L-Arginine
- Arm III - high dose (Experimental): Oral L-arginine twice daily = 6 capsules per day.
  Interventions: Drug: Oral L-Arginine

INTERVENTIONS:
Other: Placebo — Given orally
  Arms: Arm I - Placebo; Arm II - low dose
Drug: Oral L-Arginine — Given orally 3 capsules ArginMax and 3 Placebo capsules
  Other Names: ArginMax; Placebo
  Arms: Arm II - low dose; Arm III - high dose
Drug: Oral L-Arginine — Patients will take 6 capsules of ArginMax twice daily
  Other Names: ArginMax
  Arms: Arm III - high dose

SUMMARY:
RATIONALE: L-arginine supplements may improve the quality of life and erectile function in men who are prostate cancer survivors.

PURPOSE: This randomized phase II trial is studying how well L-arginine supplementation works with or without enzyme inhibitors in treating erectile function and quality of life of prostate cancer survivors previously treated with radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the "best dose" (defined as the dose that shows the greatest improvement in the erectile function domain of the International Index of Erectile Function [IIEF] after 8 weeks of therapy) of an L-arginine/Korean ginseng/gingko biloba/damiana-based supplement (L-arginine) to be used in a subsequent phase III trial in prostate cancer survivors previously treated with radiotherapy.

Secondary

* Evaluate the toxicity of treatment with L-arginine with or without phosphodiesterase-5 inhibitors.
* Estimate trial accrual, retention, adherence, and variability.
* Assess changes in quality of life (QOL) and sexual function as defined by changes in the QOL of these patients using the Expanded Prostate Cancer Index Composite, changes in the other domains of the IIEF (i.e., orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction), changes in the Sexual Encounter Profile, and changes in the percentage of "yes" (positive) responses to either of the two global efficacy questions.

OUTLINE: Patients are stratified according to age (< 65 years vs ≥ 65 years) and current use of phosphodiesterase-5 (PDE-5) inhibitors (yes vs no). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive oral placebo twice daily (total of 6 capsules per day).
* Arm II: Patients receive oral L-arginine and oral placebo twice daily (total of 3 capsules of each per day).
* Arm III: Patients receive oral L-arginine twice daily (total of 6 capsules per day).

In all arms, treatment continues for 8 weeks in the absence of unacceptable toxicity.

Patients may also receive oral sildenafil, tadalafil, or vardenafil (PDE-5 inhibitors).

Patients complete the International Index of Erectile Function and the Expanded Prostate Cancer Index Composite-26 at baseline and at weeks 4 and 8. Patients also complete the Sexual Encounter Profile Questionnaire, FACT-P, and the Global Efficacy Questionnaire at weeks 4 and 8.

ELIGIBILITY:
INCLUSION CRITERIA:

* Male prostate cancer survivor previously treated with radiotherapy and who identifies himself as concerned with sexual quality of life, including erectile dysfunction. (seed implants are eligible)
* Had successful sexual activity prior to the commencement of radiotherapy.
* Erectile dysfunction, defined as inability to achieve or maintain an erection sufficient for satisfactory sexual performance
* Interested in sexual activity and agrees to make at least one sexual intercourse attempt with a partner every week during the study.
* The usage of PDE-5 inhibitors will be voluntary and will serve as a stratification factor. Patients taking PDE-5 inhibitors must agree to assume the responsibility for the cost of PDE-5 inhibitor treatment during the protocol period (8 week period) as this is not covered in the cost of the trial.
* Patients currently taking PDE-5 inhibitors sildenafil (Viagra®, Pfizer Pharmaceuticals), tadalafil(Cialis®, Lilly ICOS, LLC), and vardenafil (Levitra®, Bayer Healthcare / Schering Plough Corp.)must agree to take the medication only as prescribed by their treating physician.
* Patients taking PDE-5 inhibitors as part of this study must be on a stable dose of drug for at least one month prior to study entry.
* Must be able to take oral medications.
* > 6 months following completion of all cancer therapy
* No evidence of prostate cancer
* Prior malignancies allowed if no evidence of recurrent disease.
* If previously taken LHRH agonist androgen suppression (e.g, Lupron, Zoladex), anti-androgen (e.g., Casodex, Eulexin, Nilandron), or estrogenic (e.g., diethylstilbestrol) agents, serum testosterone must have returned to the laboratory normal range
* No planned surgery while on protocol or for 4 weeks following completion of protocol
* Prior cystoscopy is permitted.
* Age > 18
* ECOG performance status 0/1.
* Patients must agree not to start taking an herbal product for erectile dysfunction during the eight weeks of study intervention.

EXCLUSION CRITERIA:

* No other concurrent erectile dysfunction therapies permitted (i.e. vacuum pump,cavernosal injections, and other drug therapies). Past use of these and other therapies permitted if the patient can meet the inclusion criteria above.
* No testosterone supplementation permitted.
* Use of LHRH agonist androgen suppression (e.g, Lupron, Zoladex), anti- androgen (e.g., Casodex,Eulexin, Nilandron), or estrogenic (e.g., diethylstilbestrol) agents within the last 6 months.
* Prior prostate or lower genitourinary surgery (bladder, penis, urethra, testicles)including transurethral resection of prostate (TURP). (Prior vasectomy is allowed)
* Serious cardiovascular disease (unstable angina, supraventricular arrhythmia, myocardial infarction, symptomatic congestive heart failure, cardiac arrhythmia, coronary artery bypass surgery within 6 months prior to registration).
* Hypotension (<90/50mm Hg), or uncontrolled hypertension (>170/100 mm Hg)
* Stroke or spinal cord injury within 6 months before registration.
* Patients on Persantine, heparin, Lovenox, warfarin, ginkgo biloba, Plavix, Disalcid, other blood-thinning medication or with a history of bleeding disorders will be excluded.(Aspirin < 325mg allowed)
* Current use of cimetidine, ketoconazole, itraconazole, erythromycin, or ritonavir. Major medical or psychiatric illness which, in the opinion of the investigator, would prevent completion of treatment or would interfere with follow-up.
* Current or prior use of any organic nitrate within the last 6 months (e.g., use of nitroglycerin)
* May not receive other investigational agents or devices during 30 days prior to start of study drug.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ArginMax (l-arginine, ginseng, or ginkgo biloba)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2014-02-04 (Actual); Study Completion 2014-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James J. Urbanic, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- W F Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I - Placebo | Arm II - Low Dose | Arm III - High Dose
Started | 48 | 45 | 47
Completed | 38 | 34 | 37
Not Completed | 10 | 11 | 10
Not completed — Withdrawal by Subject | 4 | 6 | 2
Not completed — Never Started | 2 | 2 | 4
Not completed — Toxicity | 1 | 3 | 2
Not completed — Multiple Reasons | 3 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I - Placebo | Arm II - Low Dose | Arm III - High Dose | Total
Number analyzed (Participants) | 48 | 45 | 47 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 13 | 40
  >=65 years | 34 | 32 | 34 | 100
Age, Continuous [Median (Full Range); unit: years] | 68 [48 to 78] | 68 [54 to 80] | 67 [53 to 80] | 68 [48 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 48 | 45 | 47 | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 45 | 43 | 45 | 133
  Unknown or Not Reported | 2 | 1 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 17 | 17 | 47
  White | 35 | 28 | 28 | 91
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 48 | 45 | 47 | 140

OUTCOME MEASURES:

1. Primary Outcome: International Index of Erectile Function (IIEF)
Description: The International Index of Erectile Function (IIEF) questionnaire consists of 15 questions, each of which is scored on a 0 to 5 or 1 to 5 scale. It is comprised of five domains, each scored as the sum of 2 to 5 questions. Erectile function is the sum of six questions with a range from 1 to 30. Higher scores indicate better functioning.
Time Frame: 8 weeks
Population: All participants providing data at any time.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I - Placebo | Arm II - Low Dose | Arm III - High Dose
Number analyzed (Participants) | 46 | 43 | 46
units on a scale | 14.62 (1.09) | 14.26 (1.13) | 11.82 (1.11)

2. Secondary Outcome: Retention
Description: Retention is the percentage of participants who complete the 8 week visit.
Time Frame: 8 weeks
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I - Placebo | Arm II - Low Dose | Arm III - High Dose
Number analyzed (Participants) | 48 | 45 | 46
percentage of participants | 79.2 [65.0 to 89.5] | 75.6 [60.5 to 87.1] | 78.7 [64.3 to 89.3]

3. Secondary Outcome: Adherence
Description: Adherence is the percentage of prescribed pills taken by the participants
Time Frame: 8 weeks
Population: Participants who returned pill diaries.
Measure: Mean (Full Range); unit: percentage of prescribed pills
Arm/Group | Arm I - Placebo | Arm II - Low Dose | Arm III - High Dose
Number analyzed (Participants) | 42 | 41 | 40
percentage of prescribed pills | 96.5 [40 to 100] | 95.0 [50 to 100] | 95.0 [36 to 100]

4. Secondary Outcome: Assessment of Quality of Life
Description: Quality of life is quantified by the Functional Assessment of Cancer Therapy - Prostate (FACT_P) questionnaire. The FACT questionnaire is comprised of four subscales - social, emotional, functional, and physical. Each subscale is obtained by summing over 6-7 items, each of which is coded on a 0 to 4 scale. Negatively worded questions are reverse scored and higher scores for each subscale indicate better HRQOL. The social, functional, and physical subscales range from 0 to 28 while the emotional subscale ranges from 0 to 24. The overall score (FACT-G) is the sum over the four subscales and ranges from 0 to 108. Patients also completed 12 questions related to prostate cancer, and the prostate subscale score is the sum of those responses (with some items reverse scored). Scores range from 0 to 48, and as with the other FACT subscales higher scores indicate better HRQOL. FACT-P is the sum of FACT-G and the prostate subscale. This questionnaire was added half-way through the study.
Time Frame: 8 weeks
Population: All participants who completed the FACT_P at any time.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I - Placebo | Arm II - Low Dose | Arm III - High Dose
Number analyzed (Participants) | 24 | 26 | 27
units on a scale | 128.54 (3.11) | 128.67 (3.08) | 127.41 (3.15)

ADVERSE EVENTS:
Time Frame: 8 weeks of treatment plus 4 weeks after treatment ends
Description: The sample size for this section was the number of participants in each arm who had post-randomization toxicity data recorded.
Arm/Group | Arm I - Placebo | Arm II - Low Dose | Arm III - High Dose
Serious Adverse Events (participants affected / at risk) | 1/41 | 1/42 | 0/42
Other Adverse Events (participants affected / at risk) | 13/41 | 16/42 | 10/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Placebo (N=41) | Arm II - Low Dose (N=42) | Arm III - High Dose (N=42)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Placebo (N=41) | Arm II - Low Dose (N=42) | Arm III - High Dose (N=42)
Agitation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Breast Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Ejaculation Disorder (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (2) | 1 (2) | 1 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestional Disorder - Other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 3 (3) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hot Flashes (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infections and Infestations - Other (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Libido Increased (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (3)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Penile Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorder - other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes